CLINICAL TRIAL: NCT01609764
Title: Physical Activity and Movement Efficiency and Quality Sleep With Increasing Age
Brief Title: Physical Activity, Sleep and Age
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maastricht University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Basic Science
Other Study IDs: NL40040.068.12
Record Dates: First submitted 2012-04-18; First posted 2012-06-01 (Estimated); Last update posted 2016-03-16 (Estimated); Status verified 2015-04

CONDITIONS: Aging; Movement Efficiency; Sleep

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Exercise (Experimental): Follows the fitness program as described in the intervention
  Interventions: Behavioral: One year fitness training
- Control (No Intervention): Will not follow any regular fitness activity during one year

INTERVENTIONS:
Behavioral: One year fitness training — Regular training schedule of moderate intensity, at 50% of heart rate reserve, as available for the specific age group in fitness centres
  Arms: Exercise

SUMMARY:
Ageing is associated with a reduction of physical activity, movement efficiency, and quality of sleep. This leads to reduced health and well being in elderly subjects. Exercise training can increase movement efficiency and quality of sleep.

Objectives:

1. Laboratory validation test of body acceleration based indexes for movement efficiency and quality of sleep;
2. Cross-sectional analysis to assess relations between these indexes and age;
3. Intervention study to assess the effect of exercise training on daily life movement efficiency and quality of sleep in ageing subjects

45 healthy human volunteers, age 50-83 yr, BMI 20-30 kg/m2 are divided in control or intervention group. Subjects that will have practiced fitness activities in the previous year, as well as pregnant or lactating women, will be excluded.

ELIGIBILITY:
Inclusion Criteria:

* Men and women
* Age between 50-85 years
* No fitness activity in the previous year, to amplify training effects on movement efficiency and quality of sleep.
* Body mass index between 20 and 30 kg/m2, obesity limits the training capacity of subjects.

Signed informed consent by the participants

Exclusion Criteria:

* Age below 50 or above 85 years;
* body mass index below 20 kg/m2 or above 30 kg/m2;
* neurologic, cardiologic or invalidating orthopaedic disease;
* pregnancy or lactation.

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2013-01; Primary Completion 2013-10 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Changes in movement efficiency | At baseline and after 1 year
  The primary objective is to identify features of body acceleration to be included in an index to assess daily life movement efficiency. Secondly, the index is related with age to quantify how ageing affects daily life movement efficiency.
  The third objective is to show the effects of regular physical activity training on this index. The expected improvement of the index would show that exercise delays the age related decrease of movement efficiency.

SECONDARY OUTCOMES:
Changes in quality sleep | At baseline and after 1 year
  The primary objective is to identify features of body acceleration to be included in one index to assess quality of sleep in daily life. Secondly, the index is related with age to quantify how ageing affects quality of sleep.
  The third objective is to show the effects of regular physical activity training on this index. The expected improvement of the index would show that exercise delays the age related decrease of quality of sleep.

CONTACTS AND LOCATIONS:
Overall Officials: Klaas R Westerterp, Professor, Principal Investigator — Maastricht University, NUTRIM, Human biology
Locations (1):
- Maastricht University, Maastricht, Limburg, Netherlands

REFERENCES:
- [Derived] Valenti G, Bonomi AG, Westerterp KR. Walking as a Contributor to Physical Activity in Healthy Older Adults: 2 Week Longitudinal Study Using Accelerometry and the Doubly Labeled Water Method. JMIR Mhealth Uhealth. 2016 Jun 7;4(2):e56. doi: 10.2196/mhealth.5445. PMID 27268471